CLINICAL TRIAL: NCT03145857
Title: A Phase I/II Study of Gallium-68 HA-DOTATATE ([68]Ga-HA-DOTATATE) in Patients With Known or Suspected Somatostatin Receptor Positive Tumours
Brief Title: A Study to Evaluate a New Way to Identify/Diagnose Tumours With Somatostatin Receptors Using [68]Ga-HA-DOTATATE and to Ensure it is Safe to Use
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-GAL-001; HREBA.CC-16-1013 (Other: Health Research Ethics Board of Alberta Cancer Committee)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
Keywords: Gallium-68; Positron Emission Tomography; 68Ga-HA-DOTATATE
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68]Ga-HA-DOTATATE (Experimental): All participants will be imaged with [68]Ga-HA-DOTATATE PET/CT or PET/MRI for uptake by somatostatin receptor positive tumours. Up to seven [68]Ga-HA-DOTATATE scans may be performed per participant, as clinically indicated.
  Interventions: Drug: [68]Ga-HA-DOTATATE

INTERVENTIONS:
Drug: [68]Ga-HA-DOTATATE — All participants will be injected with [68]Ga-HA-DOTATATE approximately 60 minutes before PET/CT or PET/MRI scan.
  Other Names: Gallium-68 high affinity-DOTATATE; Gallium-68 DOTA-3-iodo-Tyr(3)-octreotate

SUMMARY:
A [68]Ga-HA-DOTATATE PET/CT or PET/MRI scan is a nuclear medicine test used to create pictures of the whole body that will show where somatostatin receptors are found, including on tumours. Somatostatin receptors are found on most neuroendocrine tumours (NETs), and some other types of tumours. Currently at the Cross Cancer Institute, most patients with suspected somatostatin positive tumours (e.g. NETs) have an In-111 Octreotide (Octreoscan™) scan. A scientific study has shown that a scan with a similar product ([68]Ga-DOTATATE) is more accurate than an Octreoscan™. This study will look at [68]Ga-HA-DOTATATE, a product virtually identical to [68]Ga-DOTATATE.

The purpose of this study is to: 1) demonstrate the safety of [68]Ga-HA-DOTATATE; and 2) confirm that [68]Ga-HA-DOTATATE PET/CT or PET/MRI is effective at diagnosing somatostatin positive tumours.

DETAILED DESCRIPTION:
The proposed clinical trial will be a sequential Phase I/II, diagnostic imaging, controlled, open label, single site study in a broad cross-section of patients with known or suspected somatostatin receptor positive tumours. All participants will be imaged with [68]Ga-HA-DOTATATE PET/CT or PET/MRI for uptake by somatostatin receptor positive tumours. Up to seven [68]Ga-HA-DOTATATE scans may be performed per participant, as clinically indicated. A safety evaluation will be conducted on the first 10 consecutively enrolled participants (safety sub-group), consisting of vital signs, haematology and serum biochemistry profile (pre-injection and post-imaging), and an adverse event (AE) assessment (up to 24 hours) after [68]Ga-HA-DOTATATE imaging. The safety evaluation for subsequent [68]Ga-HA-DOTATATE scan visits for participants in the safety sub-group and for the remaining participants will consist of an AE assessment while in the Nuclear Medicine department. The efficacy evaluation will include [68]Ga-HA-DOTATATE scan clinical accuracy compared to standard of care CT.

ELIGIBILITY:
Inclusion Criteria:

1. Known or suspected somatostatin receptor positive tumour including, but not limited to, GNET, PNET, pulmonary NET, PRUNK NET, pheochromocytoma, paraganglioma, medullary thyroid cancer, and medulloblastoma. A standard CT obtained within 6 months of enrolment is required. A standard MRI obtained within 6 months of enrolment is optional. Additional supporting evidence obtained within 12 months of enrolment may include: other standard imaging (In-111 octreotide (Octreoscan), [18]F-FDG PET, or [18]F-FDOPA PET); histopathology from surgery or biopsy; elevated biochemical markers (including Chromogranin A, 5-HIAA, insulin, vasoactive intestinal peptide (VIP), glucagon, gastrin, metanephrines, and/or others, as clinically indicated); and/or persistent carcinoid-like symptomology highly suspicious for the presence of NET even in absence of pathologic imaging findings by anatomic criteria;
2. Eastern Cooperative Oncology Group (ECOG) Performance Scale Score ≤ 3 within 2 weeks of enrolment;
3. At least 14 years of age;
4. Able and willing to follow instructions and comply with the protocol;
5. Ability to provide written informed consent prior to participation in the study.

Exclusion Criteria:

1. Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.);
2. Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.);
3. Any additional medical condition, serious inter-current illness or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study performance or interpretation;
4. Weight exceeding the PET/CT or PET/MR scanner limit;
5. Pregnancy;
6. Allergic reaction to DOTATATE or somatostatin analogues.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1534 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2040-08 (Estimated); Study Completion 2046-08 (Estimated)

PRIMARY OUTCOMES:
Change in vital signs after first [68]Ga-HA-DOTATATE injection (safety sub-group) | Before first [68]Ga-HA-DOTATATE injection and after [68]Ga-HA-DOTATATE scan (within ~30 min)
  Vital signs are measured before first injection of [68]Ga-HA-DOTATATE and after [68]Ga-HA-DOTATATE scan and changes will be summarized.
Changes in haematology and biochemistry after first [68]Ga-HA-DOTATATE injection (safety sub-group) | Before first [68]Ga-HA-DOTATATE injection and after [68]Ga-HA-DOTATATE scan (within ~30 min)
  A blood sample is drawn before first injection of [68]Ga-HA-DOTATATE and after [68]Ga-HA-DOTATATE scan. The haematology and biochemistry parameters will be recorded and all changes will be summarized.
Number of participants with adverse events within 24 hours (safety sub-group) | Within 24 hours of [68]Ga-HA-DOTATATE scan completion
  Participants will be evaluated for AE occurrence once the [68]Ga-HA-DOTATATE has been administered for AEs occuring within 24 h of first scan.
Number of participants with adverse events | Up to 2 hours after [68]Ga-HA-DOTATATE administration
  Participants will be evaluated for AE occurrence once the [68]Ga-HA-DOTATATE has been administered for AEs occuring while in the Nuclear Medicine Department.
Correlation of [68]Ga-HA-DOTATATE scan diagnostic effectiveness with standard of care CT | Up to 6 years
  [68]Ga-HA-DOTATATE scans will be evaluated for abnormal accumulation of [68]Ga-HA-DOTATATE. The maximum Standardized Uptake Value (SUVmax) will be determined for up to 5 lesions and compared to results of baseline standard of care CT for presence/absence of each lesion. An overall assessment of the correlation between [68]Ga-HA-DOTATATE PET/CT or PET/MRI and baseline CT will be made.

SECONDARY OUTCOMES:
Evaluation of [68]Ga-HA-DOTATATE scan changes compared to baseline scan | Up to 6 years
  As applicable, follow-up [68]Ga-HA-DOTATATE scans will be evaluated for abnormal accumulation of [68]Ga-HA-DOTATATE. The maximum Standardized Uptake Value (SUVmax) will be determined for the target lesions identified at baseline and compared to the results of the baseline [68]Ga-HA-DOTATATE. An overall assessment of the correlation between the follow-up and baseline scan will be made.
Correlation of [68]Ga-HA-DOTATATE scan diagnostic effectiveness with standard of care MRI | Up to 6 years
  [68]Ga-HA-DOTATATE scans will be evaluated for abnormal accumulation of [68]Ga-HA-DOTATATE. The maximum Standardized Uptake Value (SUVmax) will be determined for up to 5 lesions and compared to results of baseline standard of care MRI, where available, for presence/absence of each lesion. An overall assessment of the correlation between [68]Ga-HA-DOTATATE PET/CT or PET/MRI and baseline MRI will made.

CONTACTS AND LOCATIONS:
Overall Officials: Todd PW McMullen, MD, PhD, FRCSC, FACS, Principal Investigator — Associate Professor of Surgery and Oncology; Director, Division of Surgical Oncology, Department of Oncology
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No